CLINICAL TRIAL: NCT00336011
Title: Studie Zur Sicherheit Von Medtronic Schrittmachern Bei Magnetresonanz-Bildgebungsverfahren an 1,5 Tesla-Systemen Study to Evaluate Safety Medtronic Pacemakers in MR Imaging at 1.5T Tesla)
Brief Title: Safety of Cardiac Pacemakers in 1.5T Tesla MRI
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Collaborators: Medtronic (Industry)
Other Study IDs: 186/02
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2006-06-12 (Estimated); Status verified 2006-01

CONDITIONS: Heart Diseases
Keywords: pacemaker; magnetic resonance imaging; safety
MeSH Terms: conditions — Heart Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: Magnetic resonance imaging

SUMMARY:
To evaluate short-term and long-term effects by MR imaging on the technical and functional status of Medtronic pacemakers.

DETAILED DESCRIPTION:
The presence of a cardiac pacemaker (PM) is currently considered an absolute contraindication to MR imaging, and most patients with PM are excluded from having MRI. In 2002 there were approximately 2.4 million patients in the US with cardiac PM, and this number is growing by 80,000 annually. A previous study has shown that MRI is indicated in 17% of all patients with pacemakers within 12 months of device placement 1, demonstrating the need for a practical and safe approach for performing MRI on PM patients.

The aim of this study is to develop a strategy for safe performance of MR imaging at 1.5T, which included exclusion of pacemaker dependent patients and those requiring imaging of the thorax, restriction of specific absorption rate (SAR) values to minimize the risk of lead heating, and PM reprogramming to avoid interference from time varying gradient fields. The safety of this approach is then evaluated in a large group of PM patients including assessment of potential myocardial thermal injury by measuring serum troponin I and pacing capture thresholds, and performing a 3-month follow-up to evaluate long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Urgent need for an MRI examination
* Presence of a Medtronic PM system manufactured between 1993 and 2004
* Stable pacemaker physical parameters

  * Battery voltage > 2.7 V
  * Battery impedance < 2000 Ohm
  * Battery estimated remaining lifetime > 6 months
  * Lead impedances 200-2000 Ohm
* Stable pacing parameters

  * Pacing capture threshold <2.5V at a pulse duration of 0.4ms
  * Sensing > 5mV
* Minimum 3 months since pacemaker and lead implantation

Exclusion Criteria:

* PM system manufacturer other than Medtronic
* History of ventricular tachycardia (VT) or ventricular fibrillation
* Unstable angina
* Myocardial infarction within the previous 3 months
* Cardiothoracic surgery within the previous 3 months
* Complete atrioventricular block
* Absolute pacemaker dependence

  * Heart rate < 40 bpm or
  * Heart rate < 60 bpm producing neurological symptoms
* Presence of an abdominal pacemaker with lead length > 70 cm
* Presence of MRI incompatible bioimplants or other MRI incompatible materials
* Request for an MR examination of the chest, including the heart, breasts and thoracic spine

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 2002-12; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Sommer, MD, Principal Investigator — University of Bonn, Department of Radiology
Locations (1):
- University of Bonn, Department of Radiology, Bonn, North Rhine-Westphalia, Germany